CLINICAL TRIAL: NCT06870604
Title: Comparison of Laparoscopic Surgery and Open Surgery for Repair of Gastric Perforation: a Multicenter, Propensity Score-matched Analysis
Brief Title: Comparison of Laparoscopic Surgery and Open Surgery for Repair of Gastric Perforation
Status: Completed | Type: Observational
Sponsor: Dong Peng (Other)
Responsible Party: Sponsor-Investigator, Dong Peng, Principal Investigator, First Affiliated Hospital of Chongqing Medical University
Organization: First Affiliated Hospital of Chongqing Medical University (Other)
Other Study IDs: ZZ2025-131-01
Record Dates: First submitted 2025-03-06; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Gastric Perforation
Keywords: gastric perforation; laparoscopic surgery; open surgery; PSM; overall complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- the gastric perforation group: patients diagnosed as gastric perforation
  Interventions: Procedure: do open surgery; Procedure: do laparoscopic surgery

INTERVENTIONS:
Procedure: do open surgery — Open surgery was performed in patients undergoing gastric perforation
Procedure: do laparoscopic surgery — Laparoscopic surgery was performed in patients undergoing gastric perforation

SUMMARY:
Gastric perforation (GP) is a penetrating lesion of the gastric wall that accounts for 10-15% of all peptic ulcer perforations, and most GP are spontaneous perforations caused by ulcer disease. Due to the presence of gastric acid, most patients often present to the emergency department with severe abdominal or chest pain due to chemical peritonitis within a few hours of perforation. Emergency physicians often quickly diagnose GP by using a chest x-ray or CT in an upright position and the patient's symptoms. Studies have shown that about 80-85% of patients with GP had subphrenic free gas visible on x-ray in the upright position.

Surgery is currently the mainstay of treatment for most GP, and almost all cases require urgent surgical repair.2 Over the past few years, laparoscopic surgery has become increasingly popular in clinical practice due to its advantages of less pain, less scarring, and early mobility out of bed, and has become the standard treatment for many elective and emergency procedures.

Since the laparoscopic study of PPU was first published by Mouret P in 1990, investigators have launched extensive discussions on the effects of laparoscopic surgery and open surgery in patients with perforated ulcers. However, to our knowledge, there are few separate discussions on GP, and the postoperative prognosis of laparoscopic surgery for patients with GP is less clear. Therefore, the aim of this multicenter, large-scale retrospective study was to compare the clinical outcomes of laparoscopic surgery and open surgery in patients with GP, to investigate whether laparoscopic surgery is safe and feasible for patients with GP, and to provide reliable evidence for surgical strategies in patients with GP.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years;
* patients diagnosed with gastric perforation.

Exclusion Criteria:

* patients with incomplete clinical data;
* laparoscopic surgery transfer to open surgery.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients diagnosed with gastric perforation
Sampling Method: Non-Probability Sample
Enrollment: 827 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
overall survival | From date of diagnosis until the date of death from any cause or or loss to follow-up, whichever came first, assessed up to 60 months.
  Overall survival (OS) was described as time from date of diagnosis until the date of death from any cause or or loss to follow-up.

IPD SHARING:
Plan to Share IPD: No
Clinical centres conducting this study are not allowed to disclose patient information and data sharing.